CLINICAL TRIAL: NCT01323998
Title: Evaluating the Treatment Patterns in Men With Benign Prostatic Hypertrophy (Marketscan Database Study)
Brief Title: Benign Prostatic Hypertrophy Treatment Patterns & Outcomes: Marketscan
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114462
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2012-02-29 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Hyperplasia
Keywords: enlarged prostate; Benign prostatic hyperplasia; alpha-blocker; 5-alpha-reductase inhibitor
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 5ARI monotherapy: Patients with BPH receiving 5ARI monotherapy
  Interventions: Drug: 5ARI
- AB monotherapy: Patients with BPH receiving AB monotherapy
  Interventions: Drug: AB
- Early combination (5ARI + AB) therapy: Patients receiving early initiation of combination therapy with a 5ARI plus AB. Early initiation defined as starting 5ARI therapy within 30 days of initiating AB therapy
  Interventions: Drug: 5ARI; Drug: AB
- Delayed combination (5ARI + AB) therapy: Patients receiving delayed initiation of combination therapy with a 5ARI plus AB. Delayed initiation defined as starting 5ARI therapy more than 30 days but less than 6 months after initiating AB therapy
  Interventions: Drug: 5ARI; Drug: AB

INTERVENTIONS:
Drug: 5ARI — Dutasteride or Finasteride
  Groups: 5ARI monotherapy; Delayed combination (5ARI + AB) therapy; Early combination (5ARI + AB) therapy
Drug: AB — Doxazosin, Prazosin, Tamsulosin, Terazosin or Alfuzosin
  Groups: AB monotherapy; Delayed combination (5ARI + AB) therapy; Early combination (5ARI + AB) therapy

SUMMARY:
This retrospective study aims to assess treatment patterns within 1 year of initiating BPH treatment, including 5-alpha-reductase inhibitor (5ARI) monotherapy, alpha-blocker (AB) monotherapy, early combination therapy, and delayed combination therapy. The MarketScan database will be utilized for this study (2000-2008)

ELIGIBILITY:
Inclusion Criteria:

* Male
* aged 50 years or older
* a diagnostic claim for BPH
* at least one prescription claim for a 5ARI or AB in the enrollment period
* continuous eligibility for 6 months prior to and 12 months after index prescription date

Exclusion Criteria:

* diagnosis of prostate or bladder cancer during the study period
* any prostate-related surgical procedure within 1 month of the index prescription date
* prescription claim for finasteride 1 mg for male pattern baldness during the study period

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients aged 50 years or older with a diagnostic claim for BPH and at least one prescription claim for a 5ARI or AB in the enrollment period
Sampling Method: Non-Probability Sample
Enrollment: 35032 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were neither recruited nor enrolled in this retrospective observational study. Data from medical records or insurance claims databases were anonymized.
Groups:
- Alpha-blocker (AB) Monotherapy: Males aged 50 and older who had a new pharmacy claim for AB monotherapy. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 milligram (mg), or a procedure code for prostate surgery
- 5 Alpha Reductase Inhibitor (5ARI) Monotherapy: Males aged 50 and older who had a new pharmacy claim for 5ARI monotherapy. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 mg, or a procedure code for prostate surgery
- AB Plus 5ARI Combination Therapy, Early 5ARI Starters: Males aged 50 and older who had a new pharmacy claim for AB and a subsequent claim for 5ARI within 30 days of the initial AB claim. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 mg, or a procedure code for prostate surgery
- AB Plus 5ARI Combination, Therapy, Delayed 5ARI Starters: Males aged 50 and older who had a new pharmacy claim for AB and a subsequent claim for 5ARI between 30 days and one year of the initial AB claim. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 mg, or a procedure code for prostate surgery
- 5ARI Plus AB Combination Therapy: Males aged 50 and older who had a new pharmacy claim for 5ARI and a subsequent claim for AB within one year of the initial 5ARI claim. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 mg, or a procedure code for prostate surgery
Period: Overall Study
Arm/Group | Alpha-blocker (AB) Monotherapy | 5 Alpha Reductase Inhibitor (5ARI) Monotherapy | AB Plus 5ARI Combination Therapy, Early 5ARI Starters | AB Plus 5ARI Combination, Therapy, Delayed 5ARI Starters | 5ARI Plus AB Combination Therapy
Started | 200631 | 18681 | 10294 | 12052 | 6735
Completed | 200631 | 18681 | 10294 | 12052 | 6735
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alpha-blocker (AB) Monotherapy: Males aged 50 and older who had a new pharmacy claim for AB monotherapy. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 mg, or a procedure code for prostate surgery
- Total: Total of all reporting groups
Arm/Group | Alpha-blocker (AB) Monotherapy | 5 Alpha Reductase Inhibitor (5ARI) Monotherapy | AB Plus 5ARI Combination Therapy, Early 5ARI Starters | AB Plus 5ARI Combination, Therapy, Delayed 5ARI Starters | 5ARI Plus AB Combination Therapy | Total
Number analyzed (Participants) | 200631 | 18681 | 10294 | 12052 | 6735 | 248393
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (10.4) | 67.6 (10.4) | 68.8 (10.3) | 68.0 (10.1) | 68.9 (10.1) | 67.4 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 200631 | 18681 | 10294 | 12052 | 6735 | 248393

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants by Treatment Cohort With and Without a Benign Prostatic Hypertrophy (BPH) Diagnosis
Description: The number of participants treated with alpha-blocker (AB) and 5a lpha reductase inhibitor (5ARI) as monotherapy or in combination reported by the presence or absence of a diagnosis code for BPH (International Classification of Disease, Ninth Revision, Clinical Modification codes: 222.2 and 600.xx). Early combination therapy was defined as the addition of 5ARI to existing AB therapy within 30 days of the initial AB pharmacy claim. Delayed combination therapy was defined as the addition of 5ARI to AB therapy after 30 day but within one year of the initial AB pharmacy claim.
Time Frame: 4 years
Population: Males aged 50 and older with a new pharmacy claim for AB, 5ARI or a combination of both. Participants were excluded if they had a diagnosis of prostate or bladder cancer, a treatment history for male-pattern baldness with finasteride 1 milligram, or a procedure code for prostate surgery.
Measure: Number; unit: participants
Arm/Group | Alpha-blocker (AB) Monotherapy | 5 Alpha Reductase Inhibitor (5ARI) Monotherapy | AB Plus 5ARI Combination Therapy, Early 5ARI Starters | AB Plus 5ARI Combination, Therapy, Delayed 5ARI Starters | 5ARI Plus AB Combination Therapy
Number analyzed (Participants) | 200631 | 18681 | 10294 | 12052 | 6735
participants
  Participants without a diagnosis code for BPH | 122307 | 9456 | 3293 | 3674 | 2625
  Participants with a diagnosis code for BPH | 78324 | 9225 | 7001 | 8378 | 4110

ADVERSE EVENTS:
Description: This was a survey of participants, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | Alpha-blocker (AB) Monotherapy | 5 Alpha Reductase Inhibitor (5ARI) Monotherapy | AB Plus 5ARI Combination Therapy, Early 5ARI Starters | AB Plus 5ARI Combination, Therapy, Delayed 5ARI Starters | 5ARI Plus AB Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.